CLINICAL TRIAL: NCT03359304
Title: Establishment of Neurofibromatosis-associated Tumours Biobank for Future Genomic-based Research Aiming at Improved Outcome Prediction
Brief Title: The Neurofibromatosis-associated Tumor Biobank
Status: Not yet recruiting | Type: Observational
Sponsor: Ren tingting (Other)
Responsible Party: Sponsor-Investigator, Ren tingting, Musculoskeletal Tumor Center, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Other Study IDs: PKU-MPNST
Record Dates: First submitted 2017-11-25; First posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Neurofibromatoses
Keywords: bone tumor
MeSH Terms: conditions — Neurofibromatoses; Bone Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The investigator will collect specimen and blood. If the investigator finds out that the sample doesn't have enough cells to be useful, the investigator may call for an additional sample.
Oversight: FDA-regulated Device: No

SUMMARY:
Neurofibromatosis-associated Tumor is very rare bone tumor. The investigator set up the biobank to ensure every patient has the chance to participate in future research

DETAILED DESCRIPTION:
Samples of blood and other stored material such as slides,frozen tissues or leftover diagnostic material.

Questionnaire information, including health history, growth and development, physical activity and family medical history information.

If patients have been diagnosed with a neurofibromatosis-associated tumor or another condition the investigator is interested in， the investigator will ask the patient to release medical record information relating to diagnosis and treatment of neurofibromatosis-associated tumor, other cancers, blood disorders, and similar conditions.

ELIGIBILITY:
Inclusion Criteria:

Proband Inclusion criteria: A diagnosis or suspected diagnosis of neurofibromatosis-associated tumor Family member inclusion criteria: Biological parents and full biological siblings of a case diagnosed with neurofibromatosis-associated tumor

Exclusion Criteria:

non-asian

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Asia
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Detected NF-1 gene expression pattern in neurofibromatosis-asociated tumor | 3 years
  To examine the neurofibromatosis type 1(NF-1) gene expression of the patients with neurofibromatosis-associated tumor

CONTACTS AND LOCATIONS:
Overall Officials: Tingting Ren, phD, Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No